CLINICAL TRIAL: NCT05582447
Title: Pilot Study- Osmotic Fragility in Red Blood Cells of Pediatric Patients With Cholestatic Liver Disease
Brief Title: Osmotic Fragility in Red Blood Cells of Pediatric Patients With Cholestatic Liver Disease
Status: Active, not recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-0310
Record Dates: First submitted 2022-10-10; First posted 2022-10-17 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Cholestasis; Red Cell Membrane and Enzyme Abnormalities
Keywords: osmotic fragility
MeSH Terms: conditions — Cholestasis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Disease Cohort: Age greater than one year old Direct bilirubin level of >2 mg/dl. No known congenital red cell membrane defect
  Interventions: Other: ektacytometry of red blood cells
- Control: Age matched to disease cohort No evidence for cholestatic liver disease No known congenital red cell membrane defect
  Interventions: Other: ektacytometry of red blood cells

INTERVENTIONS:
Other: ektacytometry of red blood cells — Evaluate red blood cell membrane mechanical characteristics by osmotic gradient ektacytometry

SUMMARY:
Objective:

The investigators propose to perform ektacytometry on 20 pediatric patients over age one with cholestatic liver diseases and a direct bilirubin level of greater than 2 gm/dl. The most common diagnoses will be extrahepatic biliary atresia, progressive familial intrahepatic cholestasis, Alagille syndrome, autoimmune hepatitis, primary sclerosing cholangitis, and parenteral nutrition-associated cholestasis. The investigators will correlate the osmotic fragility and deformability with direct bilirubin levels, serum cholesterol levels, serum bile acid levels, and vitamin E levels.

Design/Methods:

This pilot study will be a single center, prospective cross-sectional investigation of red blood cell ektacytometry in pediatric patients with extrahepatic cholestasis who are followed at Cincinnati Children's Hospital Medical Center. The study will include all participants with cholestasis regardless of the etiology in order to maximize the number of participants. While the population will be heterogeneous, the investigators will stratify participants according to diagnosis, recognizing that only a few participants may fall into each diagnostic category. Ektacytometry will be the method utilized to measure osmotic fragility and deformability of the RBC membrane. The ektacytometry of red cells from cholestatic patients will be compared to that of red cells obtained from contemporaneous age-matched controls recruited among patients without liver disease or red cell membrane defects undergoing blood sampling for evaluation of other entities including but not confined to functional abdominal pain.

DETAILED DESCRIPTION:
Primary Aim:

The primary aim is to determine if ektacytometry of red blood cells is abnormal in a population of pediatric patients over age one with cholestasis.

Secondary Aims:

The secondary aim is to ascertain the extent at which abnormalities in bilirubin levels, bile acid levels, vitamin E levels or cholesterol levels in cholestatic patients are related to changes in red blood cell ektacytometry in this patient population.

BACKGROUND Cholestatic liver disease is an umbrella term for reduced bile flow from either extrahepatic obstruction of bile ducts or faulty hepatocyte bile secretion. Cholestasis is a well-recognized cause of dyslipidemia, and are closely associated with abnormal cholesterol and phospholipid metabolism (3). Cholesterol conversion to bile acids may be impaired, and apo-lipoprotein B binding to cholesterol may be impaired, resulting in the formation of lipoprotein X which contains apo-lipoprotein C (3). The end result of dyslipidemia in cholestatic patients is hypercholesterolemia and an increased membrane cholesterol to phospholipid ratio (3).

The lack of bile entering the digestive tract can lead to increased serum cholesterol, and abnormally high red cell membrane cholesterol: phospholipid ratios, resulting in altered red cell membrane structural integrity (4,5). To test for this phenomenon in patients with extrahepatic biliary atresia, 20 pediatric patients will be tested using ektacytometry to test the deformability and osmotic fragility of red blood cells.

Ektacytometry is a diagnostic tool used to measure the deformability of red blood cells on an osmotic gradient (6). More specifically it measures deformability due to shear stress, while the RBC are suspended in an osmotic medium (6,7). It can differentiate among several blood maladies such as hereditary spherocytosis, hereditary elliptocytosis, Southeast Asian ovalocytosis, and pyropoikilocytosis that are otherwise difficult to diagnose (8). It does this by analyzing rheological behavior under constant shear stress in vitro and using photometric analysis of deformability. This is then quantified and provides a specific ektacytometry curve (Figure 1).

The ektacytometry curve will have several unique features depending on the red blood cell being analyzed. The Omin portion of the curve represents the value of the osmolality in which 50 percent of the red blood cells lyse. The Elmax is the value of the elongation index that reaches its maximum near physiologic osmolality (300 mOsm/Kg). And lastly the Ohyp, which represents the declining portion of the curve and correlates to the initial intracellular viscosity of the cell sample.

To date, ektacytometry has not been employed systematically to characterize potential red cell abnormalities in cholestatic patients. In our analysis the ektacytometry profiles of cholestatic patients will be compared to those of historical non-cholestatic age-matched controls. The degree of fragility will be correlated with serum direct bilirubin levels, serum cholesterol levels, and vitamin E levels.

STUDY DESIGN This pilot study will be a single center, prospective cross-sectional investigation into the ektacytometry of red blood cells taken from 20 cholestatic pediatric patients followed at Cincinnati Children's Hospital. Patients are seen regularly for continued follow up in the hepatology clinic. Parents of all of these patients will be asked to participate in this investigation. The investigators will also contemporaneously analyze ektacytometry of 20 age-matched controls recruited from the general GI clinics with neither cholestatic liver disease nor know red cell membrane defects.

DURATION The study is anticipated to take approximately 6-12 months to complete. This time table includes 3-6 months to recruit patients and perform the assays and another 3-6 months to analyze the data and complete a manuscript.

ELIGIBILITY:
Inclusion Criteria:

* Disease Cohort

  * Age greater than one year old
  * Direct bilirubin level of >2 mg/dl.
  * No known congenital red cell membrane defect
* Controls

  * Age matched to disease cohort
  * No evidence for cholestatic liver disease
  * No known congenital red cell membrane defect

Exclusion Criteria:

* Disease Cohort

  * Parental refusal
  * Age <1 year old.
  * Known congenital red cell membrane defect
* Controls

  * Parental refusal
  * Age <1 year old.
  * Known congenital red cell membrane defect
  * Cholestatic liver disease

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited from Cincinnati Children's Hospital hepatology and gastroenterology clinics. Pediatric patients over age one without cholestatic liver disease and pediatric patients over the age of one with cholestatic liver diseases and a direct bilirubin level of greater than 2 gm/dl.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-04-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Red blood cell osmotic fragility | 1 year
  Omin of osmotic fragility
Red blood cell deformity | 1 year
  EImax to measure deformity of red blood cells Ohyp measures index of red cell hydration
Red blood cell hydration | 1 year
  Ohyp to measure index of red cell hydration

CONTACTS AND LOCATIONS:
Overall Officials: Samuel A Kocoshis, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be available with researchers beyond those as part of the study team at Cincinnati Children's Hospital Medical Center

REFERENCES:
- [Derived] Kocoshis TS, Kalfa TA, Miethke AG, Balistreri WF, Seu KG, Slaughter CG, Singh R, Mullen M, Kocoshis SA. Red cell abnormalities characterized by ektacytometry in children with cholestasis. Pediatr Res. 2024 Mar;95(4):1035-1040. doi: 10.1038/s41390-023-02899-2. Epub 2023 Dec 1. PMID 38040987

DOCUMENTS (1):
  • Study Protocol (2018-04-05): https://cdn.clinicaltrials.gov/large-docs/47/NCT05582447/Prot_000.pdf